CLINICAL TRIAL: NCT04317807
Title: A 12-week Randomized, Double-blind, Placebo-controlled Trial Investigating the Effects of Levetiracetam in Early Psychosis
Brief Title: R33: Levetiracetam in Early Psychosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-01820
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Early Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Drug group (Active Comparator): Participants in this group will receive 500 mg of levetiracetam twice daily for 12 weeks. After 12 weeks, levetiracetam will be gradually decreased and stopped over the next 9 days. Questionnaires will be administered at each visit to examine how participants are responding to the treatment. In addition, a brain scan and cognitive testing will be performed when feasible at the beginning and the end of the study.
  Interventions: Drug: Levetiracetam Pill
- Placebo Group (Placebo Comparator): Participants in this group will receive a placebo that looks like the levetiracetam pill twice daily for 12 weeks. After 12 weeks, the levetiracetam dose will be tapered for the next 9 days. Questionnaires will be administered at each visit to examine how participants are responding to the treatment. In addition, a brain scan and cognitive testing will be performed when feasible at the beginning and the end of the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levetiracetam Pill — Levetiracetam is an anticonvulsant that is frequently used to treat epilepsy in children and adults due to its superior tolerability, ease of use and excellent safety profile. It is rapidly absorbed and rapidly crosses the blood-brain barrier. Levetiracetam does not affect metabolism of antipsychotic drugs and may normalize hippocampal hyperactivity by decreasing excessive glutamatergic and dopaminergic transmission, thereby making it an ideal agent to test the hypothesis that reducing excessive hippocampal activity may enhance treatment of early psychosis and prevent antipsychotic toxicity. Levetiracetam will be administered in 500 mg capsules twice a day.
  Other Names: Keppra
  Arms: Study Drug group
Other: Placebo — The placebo pill (sugar pill) will look just like the levetiracetam pill but does not contain levetiracetam. Placebo will be taken along with optimal antipsychotic medication selected by either the outpatient provider or the hospital staff responsible for the participant's care. Participants will be instructed to take the placebo pill twice daily for 12 weeks.
  Arms: Placebo Group

SUMMARY:
This is a 12-week study of levetiracetam added to a second generation antipsychotic in early psychosis patients who have been ill for less than 5 years and continue to experience psychotic symptoms despite at least 8 weeks of antipsychotic treatment. Levetiracetam (Keppra) is a medication approved for the treatment of epilepsy; it reduces excessive activity in the brain. This study will test the hypotheses that adding levetiracetam will improve psychotic symptoms that are unresponsive to antipsychotic treatment and will protect the brain from atrophy (volume loss). .

DETAILED DESCRIPTION:
Participants will complete screening and baseline visits before being randomized in a 2:1 ratio to levetiracetam or placebo added to the antipsychotic medication. They will complete weekly study visits for the first 4 weeks (Baseline, Weeks 2-4) and then additional visits at Week 6, 8, and 12. Participants will be studied both by assessing change in symptom severity and cognitive performance over the 12 weeks as well as using an imaging measure of hippocampal volume integrity at baseline and week 12. After completing Week 12 or decision to withdraw prematurely from the study, participants will complete a 9 day medication tapering regimen.

ELIGIBILITY:
Inclusion Criteria

* Males and females 16 to 40 years of age, inclusive, at time of informed consent
* Must have experienced a first episode of nonaffective psychosis within 5 years and exhibit current psychosis, as defined by a score of ≥ 4 on one of the following psychosis items on the BPRS: conceptual disorganization, suspiciousness, hallucinations, unusual thought content, or grandiosity, for at least 4 days per week for at least 4 weeks
* Must have a diagnosis of either schizophrenia, schizoaffective disorder or schizophreniform disorder as established by a Structured Clinical Interview for DSM-V (SCID)
* Must have taken antipsychotic medication for a minimum of 8 weeks and at a stable dose for at least 4 weeks prior to randomization
* If assigned female at birth and of childbearing potential, patients must:

  * Have a negative urine pregnancy test (all participants assigned female at birth regardless of childbearing potential will be required to submit a pregnancy test) and
  * Not be nursing or planning a pregnancy for the duration of the study through 30 days after the last dosing visit and
  * Be abstinent or willing to use a reliable method of birth control from the screening visit and continue with the same method until termination from the study

Exclusion Criteria

* Current substance abuse or dependence for substances other than nicotine and THC (i.e. alcohol, amphetamines, barbiturates)

  * A positive urine toxic screen (excluding THC, tricyclic antidepressants, or benzodiazepines (if prescribed))
  * Moderate or severe cannabis use disorder
* Diagnosis of major mood disorder or other Axis I disorder other than Schizophrenia, Schizoaffective Disorder or Schizophreniform Disorder
* Current suicidal ideation. Suicidal ideation with intent or plan (indicated by affirmative answers to items 4 or 5 of the suicidal ideation section of the baseline C-SSRS) in the 6 months prior to screening or subjects who represent a significant risk of suicide in the opinion of the Principal Investigator
* Pregnant, nursing or positive urine pregnancy test
* Significant medical or neurological illness by history or physical exam including seizure disorder, history of loss of consciousness related to head trauma or developmental disorder including mental retardation
* Renal insufficiency (if serum creatinine is greater than laboratory limits for normal, estimated creatinine clearance must be greater than 80)
* Contraindications to MRI: metal implants, pacemaker, or other metal in the body, or claustrophobia. Individuals with tattoos will be excluded from imaging if tattoos cover more than 5% of the body surface, if a tattoo is greater than 20 cm, or if the tattoo is located on the face, neck or genitals. (Individuals with a contraindication to MRI may participate in the trial but will be excluded from the elective MRI component)
* Significant history of serious violence

  * For both inpatient and outpatient subjects, a history of serious violence as assessed by the Buss-Perry Aggression Questionnaire
  * For outpatient subjects only, a score of 5 (moderately severe) or higher on the BPRS hostility item at screening or baseline

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Change in BPRS total score | Baseline visit (week 0), Week 12 visit
  The efficacy of levetiracetam 500 mg bid vs. placebo on symptoms will be measured by the BPRS total score. Brief Psychiatric Rating Scale (BPRS) is an 18-item scale that measures positive symptoms, negative symptoms, general psychopathology and affective symptoms. Individual items are scored on a seven point likert scale. The total score is the sum of responses and ranges from 18 to 126; a higher score on the BPRS items indicates increased severity of symptoms.

SECONDARY OUTCOMES:
Change in BPRS Psychosis Subscale | Baseline visit (week 0), Week 12 visit
  Brief Psychiatric Rating Scale (BPRS) is an 18-item scale that measures positive symptoms, negative symptoms, general psychopathology and affective symptoms. Individual items are scored on a seven point likert scale. The Psychosis subscale comprises 4 items of the BPRS. The total subscale score is the sum of responses and ranges from 4 to 42; a higher score indicates increased severity of symptoms.
Change in SANS Total Score | Baseline visit (week 0), Week 12 visit
  The Scale for Assessment of Negative Symptoms (SANS) will be the instrument for measurement of negative symptoms. SANS is a 19-tiem assessment; each item is rated on a scale from 0-5. The total score is the sum of the 19 individual item ratings and ranges from 0-95; higher scores indicate greater presence of negative symptoms.
Change in MATRICS Total Score | Baseline visit (week 0), Week 12 visit
  Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery is the standard tool for assessing cognitive change in trials of cognitive-enhancing agents in schizophrenia. The assessment comprises ten individual tests to produce; the scores are converted into a standardized overall composite score, with a mean of 50 and a standard deviation of 10; higher scores indicate better cognitive performance.
Change in Hippocampal Volumetric Integrity | Baseline visit (week 0), Week 12 visit
  Assessed via MRI scan.
Change in Hippocampal Cerebral Blood Flow (CBF) | Baseline visit (week 0), Week 12 visit
  CBF measured using arterial spin labeling (ASL).

CONTACTS AND LOCATIONS:
Overall Officials: Donald Goff, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to Donald.goff@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT04317807/ICF_002.pdf